CLINICAL TRIAL: NCT06470009
Title: Portable Neuromodulation Stimulator (PoNS®) Therapy for Gait and Balance Deficits in Chronic Stroke Survivors: A Randomized Controlled Trial.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helius Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMI-SA-PoNS-STK002
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Stroke Survivors

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The active Study Intervention device will deliver high-pulse stimulation and the sham Study Intervention device will deliver no-pulse stimulation although participants will be instructed to not assume being assigned an active or sham device based on whether they can feel the stimulation in the tongue or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Sham Comparator): administration of translingual neurostimulation.
  Interventions: Device: Portable Neuromodulation Stimulator (PoNS)
- Arm 2 (Active Comparator): administration of translingual neurostimulation.
  Interventions: Device: Portable Neuromodulation Stimulator (PoNS)

INTERVENTIONS:
Device: Portable Neuromodulation Stimulator (PoNS) — The PoNS device does not deliver stimulation produced by amplitude-controlled, biphasic pulses to the anterior superior surface of the tongue through gold-plated electrodes plus physical therapy.
  Other Names: PoNS Therapy
  Arms: Arm 1
Device: Portable Neuromodulation Stimulator (PoNS) — The PoNS device delivers stimulation produced by amplitude-controlled, biphasic pulses to the anterior superior surface of the tongue through gold-plated electrodes plus physical therapy.
  Other Names: PoNS Therapy
  Arms: Arm 2

SUMMARY:
Double blind, randomized, placebo controlled, interventional clinical trial investigating the efficacy and safety of PoNS therapy on improving dynamic gait and balance deficits in chronic stroke survivors.

DETAILED DESCRIPTION:
Double blind, randomized, placebo controlled, interventional clinical trial investigating the efficacy and safety of PoNS therapy on improving dynamic gait and balance deficits in chronic stroke survivors.

The Study Intervention Therapy is a therapeutic rehabilitation program that uses the PoNS device, Active or Sham, in conjunction with individualized physical exercise regimen.

The data from this prospective, double-arm, multi-site study that will enroll 40 subjects at 2-3 different clinical sites will be used to augment efficacy and safety data obtained in the RCT (which will randomize 60 subjects 1:1 into either active PoNS combined with DGB training versus DGB training with a sham device) and the OLS (which will enroll 30 subject into one active treatment arm). The totality of the proposed clinical evidence spans 3-4 sites and approximately 120 participants.

Eligible study participants will be randomized to either active PoNS ["Study Intervention"] device ["active"] or placebo PoNS ["Study Intervention"] device ["sham"]. Participants will work with a study physical therapist - trained in PoNS Therapy by HMI Medical and registered as a PoNS Trainer (Trainer).

The Trainer will prepare a DGB training exercise program appropriate to the participant's ability level and instruct on how to perform the breathing and awareness (mindfulness) training (BAT). To ensure patient's safety during rehabilitation at home, the Trainer may assign a DGB training program slightly different from the one performed in clinic.

All participants will undergo a total of twelve weeks of DGB training program combined with active or sham device's study treatment, performed both in clinic (4 weeks, Part 1), supervised by the Trainer, and at home (8 weeks, Part 2), mostly unsupervised. At the end of the treatment period, they will be asked to return to the clinic site for the follow-up visit 12 weeks after the end of the treatment period, as shown below:

Participants will receive individualized balance and gait rehabilitation protocols appropriate to their ability level and breathing and awareness (mindfulness) training. (Table 1) During the training sessions in clinic and, subsequently, during at-home training period, the trainer can adjust /flex the DGB training based on the participant's individual response to the Study Intervention Therapy (Table 1). During Part 2, the Trainer will follow-up weekly with participants in the clinic.

Table 1

Twelve weeks after completing the 12-week treatment phase of the study, participants will be required to return to the clinic for the final assessment of treatment effect. During the 12-week follow-up period (Part 3), participants will no longer utilize the Study Intervention device but will still be encouraged to continue with their physical rehabilitation program for the duration follow-up period until the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 and < 85 years of age with a diagnosis ischemic or hemorrhagic stroke at > 6 months since stroke onset event.
2. FMA-LE scores < 34 at screening with residual paresis in the lower extremity.
3. Able to walk at least 10 feet with or without assistive device.
4. FGA score < 23 at screening.
5. Montreal Cognitive Assessment 5-min (MoCA 5-min) ≥ 6
6. Able to understand, learn and apply instructions on how to operate the PoNS device and perform the rehabilitation exercise program.

Exclusion Criteria:

1. Pre-existing neurological disorders or previous stroke affecting the other hemisphere.
2. Severe arthritis or orthopedic problems that limit passive range of motion.
3. Areas of recent bleeding or open wounds; or areas that lack normal sensation on the tongue.
4. Diagnosis of dementia or mild cognitive impairment
5. Concurrent daily use of transcutaneous electric nerve stimulation (TENS) and/or other peripheral stimulation devices (i.e. Bioness®)
6. Neurostimulation therapy over the previous 6 months
7. Cancer treatment within the past year.
8. Nonremovable metal orthodontic devices.
9. Oral health problems.
10. Chronic infectious diseases.
11. Pregnancy.
12. Sensitivity to nickel, gold or copper.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoints | 12 week
  treatment - related serious adverse events (SAE) over 12 week treatment

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Synaptic Health, Calgary, Alberta
  - Neuphysio, London, Ontario
  - Neuro-Concept, Verdun, Quebec